CLINICAL TRIAL: NCT00194220
Title: Markers in Women Undergoing Infertility Treatment
Brief Title: Infertility Markers in Serum, Urine, and Follicular Fluid
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 706658; RRU011
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Infertility
Keywords: Infertility; Oxidative stress
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, Follicular Fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is only collecting specimens from current patients of PENN Fertility Care.

The purpose of this investigation is to assess if markers of oxidative stress that are known to be associated with other medical conditions can be detected in women undergoing infertility treatment and normal women of similar age. Oxidative stress may affect a woman's eggs or the follicular cells that surround and nurture them. Other markers of to be investigated include markers of cellular aging and DNA structural changes.

Presence of these markers will be compared in blood and urine samples taken during infertility treatment, and follicular fluid at the time of IVF (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50
* Infertility patients only:

  1. Women undergoing infertility treatment (with or without in-vitro fertilization) at the University of Pennsylvania's PENN Fertility Care
  2. Verified infertility diagnosis of any of the following:

     * Endometriosis (minimal or mild)
     * Endometriosis (moderate or severe)
     * Tubal factor
     * Hypogonadotrophic hypogonadism
     * Polycystic ovary syndrome
     * Diminished ovarian reserve
     * Male factor
     * Unexplained
* Healthy normal volunteers only:

  1. Not undergoing infertility treatment
  2. Not using hormonal contraception

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Post-menopausal
* Concurrent participation in investigational trial
* Other health problems which, in the opinion of the investigator, may affect participation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing In vitro fertilization at the University of Pennsylvania
Sampling Method: Non-Probability Sample
Enrollment: 1235 (Actual)
Dates: Start 2002-09; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt T Barnhart, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Reproductive Research Unit, Philadelphia, Pennsylvania, United States